CLINICAL TRIAL: NCT03940326
Title: Comparison Study of Efficacy and Safety of Levetiracetam Versus Valproate in Treatment of Idiopathic Generalized Tonic-clonic Seizures
Brief Title: Levetiracetam Versus Valproate in Idiopathic Generalized Tonic-clonic Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Assistant professor of neurology, Mazandaran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEVIGS
Record Dates: First submitted 2019-04-30; First posted 2019-05-07 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-12

CONDITIONS: Epilepsy, Idiopathic Generalized
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized | interventions — Levetiracetam; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam
- Valproate (Active Comparator)
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam with initial dose of 500 mg per 12 hours which will be increased 500 mg/week to target dose of 2000 mg/day and the dose could be increased to 3000 mg/day if seizures recurred
  Other Names: Levebel
  Arms: Levetiracetam
Drug: Valproate — Sodium valproate with initial dose of 500 mg/day which will be increased 500 mg/week to target dose of 1500 mg/day and the dose could be increased to 2000 mg/d if seizures recurred.
  Arms: Valproate

SUMMARY:
This study is an open-label, active-controlled,non-inferiority trial comparing efficacy and safety of levetiracetam versus valproate in idiopathic generalized tonic-clonic epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥16
* At least 2 unprovoked generalized tonic-clonic seizures in last 2 years with at least one in last 6 months
* Normal brain MRI or MRI without epileptogenic lesion
* Normal electroencephalography(EEG) or existence of generalized epileptiform discharges without any focal epileptiform discharges.
* Signing consent form

Exclusion Criteria:

* History of treatment by sodium valproate or levetiracetam
* History of treatment by any anti-epileptic drug in last 6 months
* Plan for pregnancy
* Using no certain contraceptive method
* History of past or current hepatic disease
* History of past or current renal disease
* History of past or current hematologic disease
* History of known psychiatric disease
* History of status epilepticus

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Tabrizi, MD, Principal Investigator — Neurology department, Mazandaran University of Medical Sciences, Sari, Iran.
Locations (1):
- Bu Ali Sina Hospital, Sari, Mazandaran, Iran

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levetiracetam | Valproate
Started | 45 | 58
Completed | 45 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | Valproate | Total
Number analyzed (Participants) | 45 | 58 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 58 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (8.1) | 29 (9.7) | 27.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 17 | 49
  Male | 13 | 41 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 58 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Iran | 45 | 58 | 103

OUTCOME MEASURES:

1. Primary Outcome: Time to First Seizure
Description: The time interval from the beginning of the study to occurrence of the first seizure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Levetiracetam | Valproate
Number analyzed (Participants) | 45 | 58
Days | 169 (6.1) | 178 (2.2)

2. Primary Outcome: Seizure Freedom Rate
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levetiracetam | Valproate
Number analyzed (Participants) | 45 | 58
Participants | 40 | 50

3. Secondary Outcome: Withdrawal Rate
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Levetiracetam | Valproate
Number analyzed (Participants) | 45 | 58
Participants | 4 | 6

4. Secondary Outcome: Time to Withdrawal
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Levetiracetam | Valproate
Number analyzed (Participants) | 45 | 58
Days | 220 (8.7) | 172 (4.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Levetiracetam | Valproate
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/45 | 2/58
Other Adverse Events (participants affected / at risk) | 17/45 | 30/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=45) | Valproate (N=58)
Rise in liver enzymes (Hepatobiliary disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=45) | Valproate (N=58)
Weight gain (Endocrine disorders) | 0 (0) | 16 (16)
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Irregularity of menstrual period (Endocrine disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3) | 3 (3)
Tiredness (General disorders) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (6)
Dizziness/vertigo (Nervous system disorders) | 6 (6) | 1 (1)
Psychiatric symptoms (Nervous system disorders) | 9 (9) | 0 (0)
Abnormal laboratory findings (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
1. The decision to choose between two arms of the study was made based on clinicians' judgment and we could not randomized or blind the study.
2. The current results are based on a 6-month follow up of patients and the results in longer follow up periods might be different.
3. The low number of patients might decrease the power of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT03940326/Prot_SAP_000.pdf